CLINICAL TRIAL: NCT02899819
Title: MecoExpo Study Protocol
Acronym: MecoExpo
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PI10-PR-BACH
Record Dates: First submitted 2016-09-05; First posted 2016-09-14 (Estimated); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Infant, Newborn
Keywords: pesticides; exposure; in utero

ARMS (1):
- meconium (Experimental): The meconium will be sampled in the first 2 days of life
  Interventions: Other: meconium

INTERVENTIONS:
Other: meconium — The meconium will be sampled in the first 2 days of life

SUMMARY:
The MecoExpo project seeks to evaluate the in utero exposure of newborns in the Picardie region to commonly used pesticides. These pesticides were selected in a pilot study (the Mecopic study) on the basis of their toxicity (effects on foetal development, endocrine perturbation, neurological toxicity and carcinogenicity) and a certain number of indicators of pesticide use and the presence of pesticide in the environment in Picardie.

These substances (or their metabolites) will be measured in the each newborn's meconium (the first faeces after birth) and each newborn's mother's hair in the Picardie region during the study period. The mother's exposure will also be assessed using a retrospective questionnaire (filled out within a few days of the delivery).

Thus, the MecoExpo project will enable the investigators to:

1. evaluate the relationships between foetal exposure (via the meconium), maternal exposure (via the hair and the questionnaire) and clinical parameters measured at birth (term, length, weight, etc.).
2. map pesticide exposure across the Picardie region.
3. create a meconium bank in Picardie (the first ever meconium bank in France).

ELIGIBILITY:
Inclusion Criteria:

* All newborns in Picardie will be eligible. Good command of the French language by a least one of the two people with responsibility for the child will be required for filling out the questionnaire.
* The mother's place of residence must have been in Picardie during the last two trimesters of pregnancy.

Exclusion Criteria:

* Newborns with foetal distress

Max Age: 2 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1020 (Actual)
Dates: Start 2011-02; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
fœtal vs mother exposure - term | Day 2
  evaluate the relationships between foetal exposure (via the meconium), maternal exposure (via the hair and the questionnaire) and term at birth
fœtal vs mother exposure - length | Day 2
  evaluate the relationships between foetal exposure (via the meconium), maternal exposure (via the hair and the questionnaire) and length at birth
fœtal vs mother exposure - weight | Day 2
  evaluate the relationships between foetal exposure (via the meconium), maternal exposure (via the hair and the questionnaire) and weight at birth

CONTACTS AND LOCATIONS:
Overall Officials: Caroline DEGUINES, MD, Principal Investigator — CHU Amiens
Locations (11):
- France (11):
  - CH Abbeville, Abbeville
  - CHU Amiens, Amiens
  - Groupe Santé Victor Pauchet, Amiens
  - CH Beauvais, Beauvais
  - CH Chauny, Chauny
  - CH Chateau-Thierry, Château-Thierry
  - Clinique Saint Come, Compiègne
  - CH Compiegne, Compiègne
  - Groupe Hospitalier Public Sud Oise, Creil
  - CH Laon, Laon
  - CH Peronne, Péronne

REFERENCES:
- [Result] Mayhoub F, Berton T, Bach V, Tack K, Deguines C, Floch-Barneaud A, Desmots S, Stephan-Blanchard E, Chardon K. Self-reported parental exposure to pesticide during pregnancy and birth outcomes: the MecoExpo cohort study. PLoS One. 2014 Jun 20;9(6):e99090. doi: 10.1371/journal.pone.0099090. eCollection 2014. PMID 24949871